CLINICAL TRIAL: NCT02547688
Title: Assessment of the Tolerability of Dry Airflow in the Nasal Cavity During Sleep
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study sponsor discontinued
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB00046727
Record Dates: First submitted 2015-09-09; First posted 2015-09-11 (Estimated); Last update posted 2017-08-08 (Actual); Status verified 2017-08

CONDITIONS: Healthy Adults

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nasal High Flow (Other): All subjects are in this group
  Interventions: Device: Nasal High Flow

INTERVENTIONS:
Device: Nasal High Flow

SUMMARY:
Preliminary data show that high flow nasal air has been shown to reduce promote heat exchange due to evaporation of nasal mucus by the air flow resulting in heat loss. It is unclear whether unidirectional nasal airflow is well tolerated in healthy individuals. The central hypothesis of this proposal is that dry high flow nasal air will be sufficiently tolerated in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women
* Able to consent
* Age ≥ 18
* BMI<30kg/m2

Exclusion Criteria:

* Previous diagnosis of obstructive sleep apnea or sleep disorder
* History of Constant Positive Airway Pressure treatment for Obstructive Sleep Apnea
* History of recurrent epistasis
* Pregnancy (self-report)
* Deviated nasal septum
* Unstable cardiovascular disease (decompensated Congestive Heart Failure, myocardial infarction or revascularization procedures, unstable arrhythmias)
* Uncontrolled hypertension with BP > 190/110
* Daytime hypoxemia with oxygen saturation<90% (measured at history and physical examination)
* Supplemental oxygen use
* Work in transportation industry as a driver or pilot.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-01; Primary Completion 2018-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Subjective Tolerability using Questionnaire | Baseline
  Participant response to nasal high flow using 7 point Likert scale

CONTACTS AND LOCATIONS:
Overall Officials: Jason Kirkness, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States